CLINICAL TRIAL: NCT04623242
Title: A Phase II/III Randomized, Double-Blind, Placebo-Controlled, Cognitive Endpoint, Multi-Center Study of Potential Disease Modifying Therapies in Individuals at Risk for and With Dominantly Inherited Alzheimer's Disease
Brief Title: Dominantly Inherited Alzheimer Network Trial: An Opportunity to Prevent Dementia. A Study of Potential Disease Modifying Treatments in Individuals at Risk for or With a Type of Early Onset Alzheimer's Disease Caused by a Genetic Mutation.
Acronym: DIAN-TU
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eli Lilly and Company (Industry); Hoffmann-La Roche (Industry); Alzheimer's Association (Other); National Institute on Aging (NIA) (NIH); Avid Radiopharmaceuticals (Industry); Accelerating Medicines Partnership (AMP) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIAN-TU-001 (gant-sola); The Alzheimer's Association (Other Grant/Funding Number: DIAN TTU-12-243040); U01AG042791 (NIH); 2013-000307-17 (EudraCT Number); R01AG046179 (NIH); REec-2014-0817 (Registry Identifier: Spanish Clinical Studies Registry); The Alzheimer's Association (Other Grant/Funding Number: DIAN-TU Tau-15-347219); GHR Foundation (Other Grant/Funding Number: File 4401); Alzheimer's Association (Other: HDE 18S84914)
Record Dates: First submitted 2020-10-14; First posted 2020-11-10 (Actual); Results first posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-08

CONDITIONS: Alzheimers Disease; Dementia; Alzheimers Disease, Familial
Keywords: Alzheimer's; Alzheimer's Disease; Dementia; Mutation; Genetic Mutation; Dominantly Inherited Alzheimer's Disease; Dominantly Inherited Alzheimer Network; Autosomal Dominant Alzheimer's Disease; Early Onset Alzheimer's Disease; DIAN; DIAN-TU; DIAN TU; DIAD
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — gantenerumab; solanezumab

STUDY DESIGN:
Intervention Model Description: Interventional
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Gantenerumab (Experimental)
  Interventions: Drug: Gantenerumab
- Solanezumab (Experimental)
  Interventions: Drug: Solanezumab
- Matching placebo (Gantenerumab) (Placebo Comparator)
  Interventions: Drug: Matching Placebo (Gantenerumab)
- Matching Placebo (Solanezumab) (Placebo Comparator)
  Interventions: Drug: Matching Placebo (Solanezumab)

INTERVENTIONS:
Drug: Gantenerumab — Subcutaneously every 4 weeks at escalating doses
  Other Names: RO4909832
  Arms: Gantenerumab
Drug: Solanezumab — Intravenous infusion every 4 weeks at escalating doses
  Other Names: LY2062430
  Arms: Solanezumab
Drug: Matching Placebo (Gantenerumab) — Subcutaneous injection of placebo every 4 weeks
  Arms: Matching placebo (Gantenerumab)
Drug: Matching Placebo (Solanezumab) — Intravenous infusion of placebo every 4 weeks
  Arms: Matching Placebo (Solanezumab)

SUMMARY:
The purpose of this study is to assess the safety, tolerability, biomarker and cognitive efficacy of investigational products in subjects who are known to have an Alzheimer's disease-causing mutation by determining if treatment with the study drug slows the rate of progression of cognitive impairment and improves disease-related biomarkers.

This is an analysis study for an MPRP: DIAN-TU-001 Master NCT01760005

DETAILED DESCRIPTION:
The mutations in presenilin 1 (PSEN1), presenilin 2 (PSEN2) and amyloid precursor protein (APP) that are associated with dominantly inherited Alzheimer's disease have very high penetrance (near 100%). This study will target individuals who are either known to have a disease-causing mutation or who are at risk for such a mutation (the child or sibling of a proband with a known mutation) and unaware of their genetic status. Because the age at onset of cognitive changes is relatively consistent within each family and with each mutation, an age at onset is determined for each affected parent or mutation. This study will enroll subjects who are either asymptomatic and are within a specific window of time of expected age at onset for their family and/or mutation or who have symptoms of mild Alzheimer's disease.

The ability to identify individuals destined to develop Alzheimer's disease (AD) within the next 10-15 years with a high degree of confidence provides a unique opportunity to assess the efficacy of therapies while individuals are asymptomatic and/or very early stages of dementia. Families with known disease-causing mutations are extremely rare and are geographically dispersed throughout the world. These constraints necessitate a specialized study design. Many of the subjects in this study will not yet have any cognitive symptoms of AD; they will be "asymptomatic" carriers of mutations that cause dominantly inherited Alzheimer's disease and would be expected to perform normally on standard cognitive and functional testing. Imaging and fluid biomarkers will be used to demonstrate that the treatment compounds have engaged their therapeutic targets. A set of cognitive measures designed to assess the very earliest and most subtle cognitive changes will be collected. Additionally, because many at-risk individuals decide not to know whether they have the disease-associated mutation or not, some of the at-risk individuals enrolled in this study will not have the disease causing mutations; they will be "mutation negative". It is important to enroll non-carrier subjects to avoid coercion (e.g., potential subjects may be pressured into genetic testing to learn their genetic status in order to be eligible for the trial). These mutation negative individuals will be assigned to the placebo group; and will not be included in the primary efficacy or futility analyses. Subjects and site study staff will remain blinded as to these individuals' active or placebo group assignment and mutation status. Thus, the study will be double blinded for placebo and for mutation status, except for mutation positive subjects who are aware of their genetic status. There may be exceptional circumstances when required by local regulation or health authorities where enrollment may be restricted to mutation carriers only but such mandates will be thoroughly documented and agreed upon by the governing regulatory agency and sponsor. Several different therapies (each referred to as a study drug arm) will be tested in order to increase the likelihood that an effective treatment will be discovered. The compounds are selected for this trial based on mechanism of action and available data on efficacy and safety profile.

The study design includes a pooled placebo group shared by all study drug arms. Mutation positive subjects will be assigned to a study drug arm and subsequently randomized within that arm in an overall 3:1 ratio to active drug:placebo. Mutation negative subjects will all receive placebo treatment. Importantly, subjects and study staff will not be blinded as to which study drug arm (gantenerumab or solanezumab) each subject has been assigned; they will be blinded as to whether subjects have been randomized to active drug or placebo. Biomarker data will be analyzed for pre-specified endpoints consistent with the drug's mechanism of action and known effects on the tested biomarkers. The primary cognitive endpoint will be the same for all study drug arms. This study is an adaptive platform based study. Interim analyses of the imaging or fluid biomarker endpoint will assess safety and whether each study drug engages its biological targets. This biomarker approach is particularly important in this study as most study subjects will be cognitively normal at baseline and most will remain cognitively normal during the first 2 years of the study. The cognitive composite is designed to assess subtle cognitive changes that may be detectable before the onset of dementia. The cognitive multivariate disease progression model (MDPM) endpoint design will allow for detection of these subtle cognitive changes.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-80 years of age
* Individuals who know they have an Alzheimer's disease-causing mutation or are unaware of their genetic status and have dominantly inherited Alzheimer's disease (DIAD) mutation in their family.
* Are within -15 to + 10 years of the predicted or actual age of cognitive symptom onset.
* Cognitively normal or with mild cognitive impairment or mild dementia, Clinical Dementia Rating (CDR) of 0-1 (inclusive)
* Fluency in DIAN-TU trial approved language and evidence of adequate premorbid intellectual functioning
* Able to undergo Magnetic Resonance Imaging (MRI), Lumbar Puncture (LP), Positron Emission Tomography (PET), and complete all study related testing and evaluations.
* For women of childbearing potential, if partner is not sterilized, subject must agree to use effective contraceptive measures (hormonal contraception, intra-uterine device, sexual abstinence, barrier method with spermicide).
* Adequate visual and auditory abilities to perform all aspects of the cognitive and functional assessments.
* Has a Study Partner who in the investigator's judgment is able to provide accurate information as to the subject's cognitive and functional abilities, who agrees to provide information at the study visits which require informant input for scale completion.

Exclusion Criteria:

* History or presence of brain MRI scans indicative of any other significant abnormality
* Alcohol or drug dependence currently or within the past 1 year
* Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, or foreign metal objects in the eyes, skin or body which would preclude MRI scan.
* History or presence of clinically significant cardiovascular disease, hepatic/renal disorders, infectious disease or immune disorder, or metabolic/endocrine disorders
* Anticoagulants except low dose (≤ 325 mg) aspirin.
* Have been exposed to a monoclonal antibody targeting beta amyloid peptide within the past six months.
* History of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years.
* Positive urine or serum pregnancy test or plans or desires to become pregnant during the course of the trial.
* Subjects unable to complete all study related testing, including implanted metal that cannot be removed for MRI scanning, required anticoagulation and pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2020-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall J Bateman, MD, Study Director — Washington University School of Medicine
Locations (25):
- United States (10):
  - University of Alabama in Birmingham, Birmingham, Alabama
  - University of California San Diego Medical Center, La Jolla, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Washington University in St. Louis, St Louis, Missouri
  - Columbia University, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - University of Washington, Seattle, Washington
- Australia (3):
  - Neuroscience Research Australia, Randwick, New South Wales
  - Mental Health Research Institute, Melbourne, Victoria
  - The McCuster Foundation of Alzheimer's Disease Research, Nedlands, Western Australia
- Canada (3):
  - UBC Hospital, Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill Center for Studies in Aging, Verdun, Quebec
- France (5):
  - CHU de Toulouse - Hôpital Purpan, Toulouse, Haute Garonne
  - Hopital Roger Salengro - CHU Lille, Lille, Nord
  - Groupe Hospitalier Pitie-Salpetriere, Paris, Paris
  - Hopital Neurologique Pierre Wertheimer, Bron, Rhone
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen, Seine Maritime
- St Vincent's University Hospital, Dublin, Ireland
- University of Puerto Rico, School of Medicine, San Juan, Puerto Rico
- Hospital Clínic I Provincial de Barcelona, Barcelona, Spain
- The National Hospital for Neurology and Neurosurgery, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to DIAN-TU trial data will follow the DIAN-TU data access policy, which complies with the guidelines established by the Collaboration for Alzheimer's Prevention [CAP REF].
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Bateman RJ, Xiong C, Benzinger TL, Fagan AM, Goate A, Fox NC, Marcus DS, Cairns NJ, Xie X, Blazey TM, Holtzman DM, Santacruz A, Buckles V, Oliver A, Moulder K, Aisen PS, Ghetti B, Klunk WE, McDade E, Martins RN, Masters CL, Mayeux R, Ringman JM, Rossor MN, Schofield PR, Sperling RA, Salloway S, Morris JC; Dominantly Inherited Alzheimer Network. Clinical and biomarker changes in dominantly inherited Alzheimer's disease. N Engl J Med. 2012 Aug 30;367(9):795-804. doi: 10.1056/NEJMoa1202753. Epub 2012 Jul 11. PMID 22784036
- [Background] Farlow M, Arnold SE, van Dyck CH, Aisen PS, Snider BJ, Porsteinsson AP, Friedrich S, Dean RA, Gonzales C, Sethuraman G, DeMattos RB, Mohs R, Paul SM, Siemers ER. Safety and biomarker effects of solanezumab in patients with Alzheimer's disease. Alzheimers Dement. 2012 Jul;8(4):261-71. doi: 10.1016/j.jalz.2011.09.224. Epub 2012 Jun 5. PMID 22672770
- [Background] Bateman RJ, Benzinger TL, Berry S, Clifford DB, Duggan C, Fagan AM, Fanning K, Farlow MR, Hassenstab J, McDade EM, Mills S, Paumier K, Quintana M, Salloway SP, Santacruz A, Schneider LS, Wang G, Xiong C; DIAN-TU Pharma Consortium for the Dominantly Inherited Alzheimer Network. The DIAN-TU Next Generation Alzheimer's prevention trial: Adaptive design and disease progression model. Alzheimers Dement. 2017 Jan;13(1):8-19. doi: 10.1016/j.jalz.2016.07.005. Epub 2016 Aug 29. PMID 27583651
- [Background] Mills SM, Mallmann J, Santacruz AM, Fuqua A, Carril M, Aisen PS, Althage MC, Belyew S, Benzinger TL, Brooks WS, Buckles VD, Cairns NJ, Clifford D, Danek A, Fagan AM, Farlow M, Fox N, Ghetti B, Goate AM, Heinrichs D, Hornbeck R, Jack C, Jucker M, Klunk WE, Marcus DS, Martins RN, Masters CM, Mayeux R, McDade E, Morris JC, Oliver A, Ringman JM, Rossor MN, Salloway S, Schofield PR, Snider J, Snyder P, Sperling RA, Stewart C, Thomas RG, Xiong C, Bateman RJ. Preclinical trials in autosomal dominant AD: implementation of the DIAN-TU trial. Rev Neurol (Paris). 2013 Oct;169(10):737-43. doi: 10.1016/j.neurol.2013.07.017. Epub 2013 Sep 6. PMID 24016464
- [Background] Wang G, Berry S, Xiong C, Hassenstab J, Quintana M, McDade EM, Delmar P, Vestrucci M, Sethuraman G, Bateman RJ; Dominantly Inherited Alzheimer Network Trials Unit. A novel cognitive disease progression model for clinical trials in autosomal-dominant Alzheimer's disease. Stat Med. 2018 Sep 20;37(21):3047-3055. doi: 10.1002/sim.7811. Epub 2018 May 14. PMID 29761523
- [Background] Weninger S, Carrillo MC, Dunn B, Aisen PS, Bateman RJ, Kotz JD, Langbaum JB, Mills SL, Reiman EM, Sperling R, Santacruz AM, Tariot PN, Welsh-Bohmer KA. Collaboration for Alzheimer's Prevention: Principles to guide data and sample sharing in preclinical Alzheimer's disease trials. Alzheimers Dement. 2016 May;12(5):631-2. doi: 10.1016/j.jalz.2016.04.001. No abstract available. PMID 27157073
- [Background] Grill JD, Bateman RJ, Buckles V, Oliver A, Morris JC, Masters CL, Klunk WE, Ringman JM; Dominantly Inherited Alzheimer's Network. A survey of attitudes toward clinical trials and genetic disclosure in autosomal dominant Alzheimer's disease. Alzheimers Res Ther. 2015 Jul 22;7(1):50. doi: 10.1186/s13195-015-0135-0. eCollection 2015. PMID 26203303
- [Background] McDade E, Bateman RJ. Stop Alzheimer's before it starts. Nature. 2017 Jul 12;547(7662):153-155. doi: 10.1038/547153a. No abstract available. PMID 28703214
- [Background] McDade E, Wang G, Gordon BA, Hassenstab J, Benzinger TLS, Buckles V, Fagan AM, Holtzman DM, Cairns NJ, Goate AM, Marcus DS, Morris JC, Paumier K, Xiong C, Allegri R, Berman SB, Klunk W, Noble J, Ringman J, Ghetti B, Farlow M, Sperling RA, Chhatwal J, Salloway S, Graff-Radford NR, Schofield PR, Masters C, Rossor MN, Fox NC, Levin J, Jucker M, Bateman RJ; Dominantly Inherited Alzheimer Network. Longitudinal cognitive and biomarker changes in dominantly inherited Alzheimer disease. Neurology. 2018 Oct 2;91(14):e1295-e1306. doi: 10.1212/WNL.0000000000006277. Epub 2018 Sep 14. PMID 30217935
- [Background] Ryman DC, Acosta-Baena N, Aisen PS, Bird T, Danek A, Fox NC, Goate A, Frommelt P, Ghetti B, Langbaum JB, Lopera F, Martins R, Masters CL, Mayeux RP, McDade E, Moreno S, Reiman EM, Ringman JM, Salloway S, Schofield PR, Sperling R, Tariot PN, Xiong C, Morris JC, Bateman RJ; Dominantly Inherited Alzheimer Network. Symptom onset in autosomal dominant Alzheimer disease: a systematic review and meta-analysis. Neurology. 2014 Jul 15;83(3):253-60. doi: 10.1212/WNL.0000000000000596. Epub 2014 Jun 13. PMID 24928124
- [Background] Weng H, Bateman R, Morris JC, Xiong C. Validity and power of minimization algorithm in longitudinal analysis of clinical trials. Biostat Epidemiol. 2017;1(1):59-77. doi: 10.1080/24709360.2017.1331822. Epub 2017 Jun 13. PMID 29250611
- [Derived] Wagemann O, Liu H, Wang G, Shi X, Bittner T, Scelsi MA, Farlow MR, Clifford DB, Supnet-Bell C, Santacruz AM, Aschenbrenner AJ, Hassenstab JJ, Benzinger TLS, Gordon BA, Coalier KA, Cruchaga C, Ibanez L, Perrin RJ, Xiong C, Li Y, Morris JC, Lah JJ, Berman SB, Roberson ED, van Dyck CH, Galasko D, Gauthier S, Hsiung GR, Brooks WS, Pariente J, Mummery CJ, Day GS, Ringman JM, Mendez PC, St George-Hyslop P, Fox NC, Suzuki K, Okhravi HR, Chhatwal J, Levin J, Jucker M, Sims JR, Holdridge KC, Proctor NK, Yaari R, Andersen SW, Mancini M, Llibre-Guerra J, Bateman RJ, McDade E; Dominantly Inherited Alzheimer Network-Trials Unit. Downstream Biomarker Effects of Gantenerumab or Solanezumab in Dominantly Inherited Alzheimer Disease: The DIAN-TU-001 Randomized Clinical Trial. JAMA Neurol. 2024 Jun 1;81(6):582-593. doi: 10.1001/jamaneurol.2024.0991. PMID 38683602
- [Derived] Atkins KJ, Evered L, Scott DA, Fowler C, Masters CL, Silbert B. Cerebrospinal fluid sampling for research of Alzheimer's disease and other neurodegenerative diseases when lumbar punctures are performed by anaesthetists. BMJ Neurol Open. 2022 Sep 5;4(2):e000335. doi: 10.1136/bmjno-2022-000335. eCollection 2022. PMID 36110925
- See also: Expanded registry — http://www.dianexr.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study assigned treatment to 194 participants, 1 participant enrolled in the solanezumab arm did not receive treatment. Of the 193 participants, there were 144 mutation positive participants who were treated. Two of these participants did not have post-baseline data and were excluded from the MITT. Forty-nine mutation negative participants were enrolled across the 2 drug arms but are not part of the analysis population.
Pre-assignment Details: Primary analyses used a pooled control group (gantenerumab and solanezumab shared, mutation positive placebo with dynamic borrowing of DIAN-OBS data).
Groups:
- Gantenerumab: Gantenerumab: Subcutaneously every 4 weeks at escalating doses
  Participants randomized to gantenerumab were then randomized to either active drug or placebo at a 3:1 ratio. All mutation negative participants were assigned to placebo.
  For analysis purposes, mutation positive placebos were pooled for outcome measures.
- Solanezumab: Solanezumab: Intravenous infusion every 4 weeks at escalating doses
  Participants randomized to solanezumab were then randomized to either active drug or placebo at a 3:1 ratio. All mutation negative participants were assigned to placebo.
  For analysis purposes, mutation positive placebos were pooled for outcome measures. Some secondary measures used direct placebo as specified in the respective outcomes (those randomized to solanezumab only)
- Mutation Positive Placebo: Mutation positive placebos enrolled under each arm but pooled for result reporting.
- Mutation Negative Placebo: Mutation negative participants receiving placebo. Not analyzed as part of the Pooled Placebo Group; analyzed for safety.
- DIAN-OBS: Participants from the DIAN Observational study meeting specific criteria as outlined in the posted Statistical Analysis Plan.
Period: Overall Study
Arm/Group | Gantenerumab | Solanezumab | Mutation Positive Placebo | Mutation Negative Placebo | DIAN-OBS
Started | 52 | 52 | 40 | 49 | 69
Completed | 39 | 36 | 30 | 26 | 69
Not Completed | 13 | 16 | 10 | 23 | 0
Not completed — Withdrawal by Subject | 7 | 12 | 5 | 7 | 0
Not completed — Reason Not Disclosed to protect treatment and genetic unblinding | 6 | 4 | 5 | 3 | 0
Not completed — Subject unblinded to mutation status | 0 | 0 | 0 | 13 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics relative to the primary endpoint measures do not include mutation negative placebos because the primary analysis is only run on the MITT population which excludes mutation negative.
Groups:
- Mutation Negative Placebo: Mutation Negative Placebos enrolled under each arm but pooled for this reporting.
- DIAN-OBS Control Group: Data from participants in the DIAN-OBS study who met DIAN-TU inclusion criteria were used as natural history controls for improved estimates of the placebo group.
- Total: Total of all reporting groups
Arm/Group | Gantenerumab | Solanezumab | Mutation Positive Placebo | Mutation Negative Placebo | DIAN-OBS Control Group | Total
Number analyzed (Participants) | 52 | 52 | 40 | 49 | 69 | 262
Age, Continuous [Mean (Standard Deviation); unit: years] — Represents Age at randomization (DIAN-TU-001) or age at first visit meeting inclusion criteria for DIAN-TU-001 analysis (DIAN-OBS) Population: Measure Analysis Population Description: Fifty-two participants were randomized to the solanezumab arm; two did not have post-baseline data and were excluded from the modified intent-to-treat population.
  years
    number analyzed (Participants) | 52 | 50 | 40 | 49 | 69 | 260
    (all) | 46 (10.8) | 42.7 (9.6) | 44.2 (9.6) | 42.6 (9.3) | 42.3 (9.6) | 43.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Fifty-two participants were randomized to the solanezumab arm; two did not have post-baseline data and were excluded from the modified intent-to-treat population.
  Participants
    number analyzed (Participants) | 52 | 50 | 40 | 49 | 69 | 260
    Female | 21 | 29 | 22 | 23 | 47 | 142
    Male | 31 | 21 | 18 | 26 | 22 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Fifty-two participants were randomized to the solanezumab arm; two did not have post-baseline data and were excluded from the modified intent-to-treat population.
  Participants
    number analyzed (Participants) | 52 | 50 | 40 | 49 | 69 | 260
    Hispanic or Latino | 7 | 7 | 5 | 11 | 15 | 45
    Not Hispanic or Latino | 45 | 43 | 35 | 38 | 53 | 214
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants] — Population: Measure Analysis Population Description: Fifty-two participants were randomized to the solanezumab arm; two did not have post-baseline data and were excluded from the modified intent-to-treat population.
  participants
    Canada: number analyzed (Participants) | 52 | 50 | 40 | 49 | 69 | 260
    Canada | 4 | 3 | 5 | 4 | 0 | 16
    United States: number analyzed (Participants) | 52 | 50 | 40 | 49 | 69 | 260
    United States | 32 | 30 | 18 | 35 | 35 | 150
    United Kingdom: number analyzed (Participants) | 52 | 50 | 40 | 49 | 69 | 260
    United Kingdom | 5 | 5 | 4 | 2 | 5 | 21
    Australia: number analyzed (Participants) | 52 | 50 | 40 | 49 | 69 | 260
    Australia | 4 | 6 | 5 | 1 | 12 | 28
    France: number analyzed (Participants) | 52 | 50 | 40 | 49 | 69 | 260
    France | 4 | 5 | 4 | 7 | 0 | 20
    Spain: number analyzed (Participants) | 52 | 50 | 40 | 49 | 69 | 260
    Spain | 3 | 1 | 4 | 0 | 0 | 8
    Argentina: number analyzed (Participants) | 0 | 0 | 0 | 0 | 69 | 69
    Argentina |  |  |  |  | 4 | 4
    Japan: number analyzed (Participants) | 0 | 0 | 0 | 0 | 69 | 69
    Japan |  |  |  |  | 3 | 3
    Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 69 | 69
    Germany |  |  |  |  | 10 | 10
APOE4 [Count of Participants; unit: Participants] — APOE refers to presence of at least one ε4 allele of apolipoprotein E Population: APOE was not included for the external DIAN-OBS Control Group because the data was not available from a CLIA certified lab
  Participants
    number analyzed (Participants) | 52 | 50 | 40 | 49 | 0 | 191
    (all) | 16 | 14 | 13 | 16 |  | 59
Enrollment EYO [Mean (Standard Deviation); unit: years] — EYO represents the estimated years to symptom onset as recorded by the investigator.
  This EYO is determined based on family history and clinician assessment to determine EYO eligibility for the DIAN-TU-001 trial, and no such assessment was done within DIAN-OBS as there was no EYO requirement for entry. Population: Fifty-two participants were randomized to the solanezumab arm; two did not have post-baseline data and were excluded from the modified intent-to-treat population. Data could not be reported for the DIAN-Obs Control group for the International Shopping List Test-Delayed Recall (ISLT) because data was not collected.
  years
    number analyzed (Participants) | 52 | 50 | 40 | 49 | 0 | 191
    (all) | -3.5 (7.1) | -2.4 (7.1) | -3.5 (7.6) | -4.8 (6.41) |  | -3.25 (7.2)
Digit Symbol Substitution Test [Mean (Standard Deviation); unit: score on a scale] — Digit Symbol is a subtest of the Wechsler Adult Intelligence Scale (WAIS-R). This test engages multiple cognitive abilities, including attention, psychomotor speed, complex scanning, visual tracking, and immediate memory.
  Scores range from 0 to 93, with lower scores indicating poorer cognitive performance Population: Fifty-two participants were randomized to the solanezumab arm; two did not have post-baseline data and were excluded from the modified intent-to-treat population. DIAN Obs control group only analyzed 68 participants as one participant did not have a baseline measure.
  score on a scale
    number analyzed (Participants) | 52 | 50 | 40 | 49 | 68 | 259
    (all) | 46.96 (20.56) | 46.06 (19.94) | 46.63 (19.12) | 60.78 (13.01) | 50.34 (18.57) | 47.76 (19.45)
MMSE [Mean (Standard Deviation); unit: score on a scale] — Mini Mental State Exam is a 30-point test used to measure thinking ability (or "cognitive impairment").
  The test measures the following:
  * orientation to time and place (knowing where you are, and the season or day of the week)
  * short-term memory (recall)
  * attention and ability to solve problems (like spelling a simple word backwards)
  * language (identifying common objects by name)
  * comprehension and motor skills (drawing a slightly complicated shape like two pentagons intersecting)
  Scores range from 0 to 30, with lower scores indicating poorer cognitive performance. Population: Fifty-two participants were randomized to the solanezumab arm; two did not have post-baseline data and were excluded from the modified intent-to-treat population. DIAN Obs control group only analyzed 68 participants as one participant did not have a baseline measure.
  score on a scale
    number analyzed (Participants) | 52 | 50 | 40 | 49 | 68 | 259
    (all) | 27.10 (3.45) | 26.72 (4.11) | 26.68 (3.97) | 29.08 (1.17) | 26.96 (3.22) | 26.88 (3.63)
Logical Memory Delayed Recall Test [Mean (Standard Deviation); unit: score on a scale] — Subtest of the Wechsler Memory Scale-Revised Standardized assessment of narrative episodic memory. A short story is orally presented and approximately 20 or 30 min later, examinee is asked to recall the story (delayed recall).
  Scores range from 0 to 25, with lower scores indicating poorer cognitive performance Population: Fifty-two participants were randomized to the solanezumab arm; two did not have post-baseline data and were excluded from the modified intent-to-treat population. Only 51 analyzed for this measure in the gantenerumab as 1 participant did not have a baseline measure.
  score on a scale
    number analyzed (Participants) | 51 | 50 | 40 | 49 | 69 | 259
    (all) | 9.9 (6.33) | 9.86 (6.86) | 9.4 (6.45) | 14.55 (3.72) | 9.32 (6.42) | 9.60 (6.47)
International Shopping List Test-Delayed Recall (ISLT) [Mean (Standard Deviation); unit: score on a scale] — International Shopping List Task-Delayed Recall (ISLT) is a classic list-learning test that measures verbal learning & memory.
  Scores range from 0 to 12, with lower scores indicating poorer cognitive performance. Population: Fifty-two participants were randomized to the solanezumab arm; two did not have post-baseline data and were excluded from the modified intent-to-treat population. Only 51 analyzed here for gantenerumab as 1 participant did not have a baseline measure.
  score on a scale
    number analyzed (Participants) | 51 | 50 | 40 | 49 | 0 | 190
    (all) | 5.96 (4.04) | 6.56 (3.95) | 5.80 (4.42) | 8.80 (1.99) |  | 6.13 (4.10)

OUTCOME MEASURES:

1. Primary Outcome: Assess Cognitive Efficacy in Individuals With Mutations Causing Dominantly Inherited AD as Measured by the DIAN-Multivariate Cognitive Endpoint (DIAN-MCE);
Description: Multivariate Disease Progression Model adjusted for Estimated Years to Onset (EYO)and includes all timepoints up to treatment discontinuation. The treatment effect is reported relative to the mutation positive placebo arm.
  Multivariate Cognitive Endpoint comprising: (i) Wechsler Memory Scale-Revised Logical Memory Delayed Recall Test (MEMUNITS), (ii) Wechsler Adult Intelligence Scale Digit Symbol Substitution Test (WAIS), (iii) Mini-Mental State Examination (MMSE), and (iv) International Shopping List Task (ISLT). Measurements for each test were normalized using the mean (SD) at DIAN-TU-001 baseline for mutation negative subjects. Higher scores indicate more favourable cognitive performance.
Time Frame: Baseline through Week 260
Population: The endpoint itself is a ratio based on feeding z-scores for four separate parameters into a model, with programming providing the ratio under model assumptions rather than providing a treatment-specific value this is used to generate the ratio. The four individual parameters are described in other outcomes. There are no "by-arm" values for any MDPM analysis.
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Gantenerumab vs. Mutation Positive Placebo: Gantenerumab: Subcutaneously every 4 weeks at escalating doses; Matching Placebo
- Solanezumab vs. Mutation Positive Placebo: Solanezumab: Intravenous infusion every 4 weeks at escalating doses; Matching Placebo
Arm/Group | Gantenerumab vs. Mutation Positive Placebo | Solanezumab vs. Mutation Positive Placebo
Number analyzed (Participants) | 161 | 160
Ratio | 1.063 (0.059) | 1.255 (0.061)
Statistical Analysis 1: Comparison: Gantenerumab vs. Mutation Positive Placebo; Test type: Superiority; A priori threshold for statistical significance; Ratio = 1.063, Standard Deviation 0.059
Statistical Analysis 2: Comparison: Solanezumab vs. Mutation Positive Placebo; Test type: Superiority; A priori threshold for statistical significance; Ratio = 1.255, Standard Deviation 0.061

2. Secondary Outcome: Gantenerumab: Rate of Change Over Time- Clinical Dementia Rating Sum of Boxes (CDR-SB)
Description: CDR-SB score is considered a more detailed quantitative general index of cognition and function, and provides more information than the global CDR score in patients with mild dementia
  Scores range from 0-18 with lower scores showing more favorable cognitive function.
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: Number analyzed represents actual data collections at each collection time point. Data unavailable at any time point was not collected for various reasons i.e. participant attrition or common close design (participants did not reach that time point before trial end).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Mutation Positive Placebos: Mutation positive placebos enrolled under each arm but pooled for result reporting.
Arm/Group | Gantenerumab | Mutation Positive Placebos
Number analyzed (Participants) | 52 | 40
units on a scale
  Week 52 | 0.74 (0.202) | 0.44 (0.231)
  Week 104: number analyzed (Participants) | 46 | 36
  Week 104 | 1.27 (0.364) | 1.36 (0.414)
  Week 156: number analyzed (Participants) | 41 | 32
  Week 156 | 1.95 (0.511) | 2.28 (0.580)
  Week 208: number analyzed (Participants) | 36 | 30
  Week 208 | 2.96 (0.726) | 3.24 (0.819)
  Week 260: number analyzed (Participants) | 13 | 7
  Week 260 | 4.61 (1.220) | 5.76 (1.437)
Statistical Analysis 1: Comparison: Gantenerumab vs Mutation Positive Placebos; Test type: Other; p = 0.805, t-test, 2 sided; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-2.46 to 1.92], Standard Error of Mean 1.094

3. Secondary Outcome: Gantenerumab: Rate of Change Over Time- Functional Assessment Scale (FAS)
Description: The Functional Assessment Scale is to be administered and completed by the study partner about subjects for whom they care. This scale measures instrumental activities of daily living such as preparing balanced meals and managing personal finances. The intent of the FAS is to assess change in an individual's functional activities, relative to previously attained abilities, that are caused by cognitive dysfunction. If the study partner indicates that the subject no longer performs a particular task, it is reasonable to probe further and ask if they think the subject could still do the task. This will help tease out the relevant cognitive impairment
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Gantenerumab | Mutation Positive Placebos
Number analyzed (Participants) | 52 | 40
units on a scale
  Week 52: number analyzed (Participants) | 48 | 36
  Week 52 | 1.23 (0.408) | 1.40 (0.469)
  Week 104: number analyzed (Participants) | 42 | 31
  Week 104 | 2.34 (0.680) | 2.44 (0.790)
  Week 156: number analyzed (Participants) | 37 | 29
  Week 156 | 3.45 (0.921) | 4.07 (1.061)
  Week 208: number analyzed (Participants) | 34 | 27
  Week 208 | 4.34 (1.202) | 5.55 (1.373)
  Week 260: number analyzed (Participants) | 13 | 7
  Week 260 | 6.40 (1.730) | 5.69 (2.073)
Statistical Analysis 1: Comparison: Gantenerumab vs Mutation Positive Placebos; Test of equality (any treatment difference); Test type: Other; p = 0.512, t-test, 2 sided; Mean Difference (Final Values) = -1.20, 95% CI 2-sided [-4.83 to 2.43], Standard Error of Mean 1.823

4. Secondary Outcome: Gantenerumab: Imaging Measures Composite [11C] PiB Partial Volume Corrected Regional Spread Function Standardized Uptake Value Ratio - Composite
Description: In vivo quantification of β-amyloid deposition using positron emission tomography. This measure is a composite of brain regions. Higher scores indicate worse disease stage.
Time Frame: Baseline, Weeks 52, 104 and 208
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Gantenerumab | Mutation Positive Placebos
Number analyzed (Participants) | 52 | 40
Ratio
  Week 52: number analyzed (Participants) | 47 | 37
  Week 52 | -0.006 (0.0402) | 0.103 (0.0454)
  Week 104: number analyzed (Participants) | 40 | 33
  Week 104 | -0.106 (0.0422) | 0.134 (0.0470)
  Week 208: number analyzed (Participants) | 33 | 25
  Week 208 | -0.334 (0.0736) | 0.306 (0.0839)
Statistical Analysis 1: Comparison: Gantenerumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p < 0.001, t-test, 2 sided; Median Difference (Final Values) = -0.641, 95% CI 2-sided [-0.864 to -0.417], Standard Error of Mean 0.1115

5. Secondary Outcome: Solanezumab: Clinical Measures- Clinical Dementia Rating (CDR)
Description: Clinical Dementia Rating - Global Score - Number of Subjects with an Increase from Baseline by Visit
Time Frame: Baseline and Weeks 52, 104, 156, and 208
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
Participants
  Week 52: number analyzed (Participants) | 49 | 40
  Week 52: Increase from baseline CDR Global Score | 11 | 8
  Week 52: No increase from baseline CDR Global Score | 38 | 32
  Week 104: number analyzed (Participants) | 47 | 36
  Week 104: Increase from baseline CDR Global Score | 18 | 8
  Week 104: No increase from baseline CDR Global Score | 29 | 28
  Week 156: number analyzed (Participants) | 42 | 32
  Week 156: Increase from baseline CDR Global Score | 16 | 13
  Week 156: No increase from baseline CDR Global Score | 26 | 19
  Week 208: number analyzed (Participants) | 36 | 30
  Week 208: Increase from baseline CDR Global Score | 12 | 8
  Week 208: No increase from baseline CDR Global Score | 24 | 22
  Week 260: number analyzed (Participants) | 13 | 7
  Week 260: Increase from baseline CDR Global Score | 5 | 3
  Week 260: No increase from baseline CDR Global Score | 8 | 4
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any difference in the proportion of increase in the endpoint); p = 0.5573, Chi-squared; Ratio = 0.3443

6. Secondary Outcome: Solanezumab: Clinical Measures- CDR Sum of Boxes (CDR-SB)
Description: CDR-SB score is considered a more detailed quantitative general index and provides more information than the global CDR score in patients with mild dementia
  Scores range from 0-18 with lower scores showing more favorable cognitive function.
Time Frame: Baseline and Weeks 52, 104, 156, and 208
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
units on a scale
  Week 52: number analyzed (Participants) | 49 | 40
  Week 52 | 0.90 (0.208) | 0.44 (0.231)
  Week 104: number analyzed (Participants) | 47 | 36
  Week 104 | 1.87 (0.367) | 1.36 (0.414)
  Week 156: number analyzed (Participants) | 42 | 32
  Week 156 | 2.55 (0.512) | 2.28 (0.580)
  Week 208: number analyzed (Participants) | 36 | 30
  Week 208 | 3.65 (0.723) | 3.24 (0.819)
  Week 260: number analyzed (Participants) | 13 | 7
  Week 260 | 4.87 (1.212) | 5.76 (1.437)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.707, t-test, 2 sided; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-1.77 to 2.60], Standard Error of Mean 1.092

7. Secondary Outcome: Solanezumab: Clinical Measures- Geriatric Depression Scale (GDS)
Description: The Geriatric Depression Scale (GDS) is a self-report measure of depression in older adults. Users respond in a "Yes/No" format. Of the 15 items, 10 indicate the presence of depression when answered positively while the other 5 are indicative of depression when answered negatively.
  Scores range from 0-15 for completed questionnaires. A score of 88 is recorded for participants unable to complete the test.
  Lower scores show more favorable outcome.
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
score on a scale
  Week 52: number analyzed (Participants) | 49 | 40
  Week 52 | 0.20 (0.230) | -0.14 (0.255)
  Week 104: number analyzed (Participants) | 47 | 35
  Week 104 | 0.06 (0.265) | 0.03 (0.304)
  Week 156: number analyzed (Participants) | 39 | 32
  Week 156 | -0.22 (0.250) | -0.07 (0.276)
  Week 208: number analyzed (Participants) | 35 | 28
  Week 208 | -0.12 (0.294) | 0.36 (0.328)
  Week 260: number analyzed (Participants) | 13 | 6
  Week 260 | -0.16 (0.544) | 0.66 (0.820)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.283, t-test, 2 sided; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-1.35 to 0.40], Standard Error of Mean 0.440

8. Secondary Outcome: Solanezumab: Clinical Measures- Neuropsychiatric Inventory Questionnaire (NPI-Q)
Description: The questionnaire is to be administered and completed by the study partner about patients for whom they care. Each of the 12 NPI-Q domains contains a survey question that reflects cardinal symptoms of that domain. Initial responses to each domain question are "Yes"(present) or "No" (absent). If the response to the domain question is "No", the study partner goes to the next question. If "Yes", the study partner then rates both the Severity of the symptoms present within the last month on a 3-point scale and the associated impact of the symptom manifestations on them (i.e. Caregiver Distress) using a 5-point scale. The NPI-Q provides symptom 'Severity' and 'Distress' ratings for each symptom reported, and total 'Severity' and 'Distress' scores reflecting the sum of individual domain scores.
  Scores range from 0-36 with lower scores indicating more favorable cognitive function.
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
score on a scale
  Week 52: number analyzed (Participants) | 49 | 40
  Week 52 | 0.49 (0.416) | 1.06 (0.460)
  Week 104: number analyzed (Participants) | 47 | 35
  Week 104 | 0.70 (0.463) | 1.54 (0.530)
  Week 156: number analyzed (Participants) | 42 | 32
  Week 156 | 1.31 (0.459) | 1.10 (0.522)
  Week 208: number analyzed (Participants) | 36 | 30
  Week 208 | 2.11 (0.575) | 1.74 (0.639)
  Week 260: number analyzed (Participants) | 13 | 7
  Week 260 | 1.83 (0.934) | 1.16 (1.212)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.674, t-test, 2 sided; Mean Difference (Final Values) = 0.36, 95% CI 2-sided [-1.34 to 2.07], Standard Error of Mean 0.859

9. Secondary Outcome: Solanezumab: Clinical Measures- Functional Assessment Scale (FAS)
Description: The Functional Assessment Scale is to be administered and completed by the study partner about subjects for whom they care. This scale measures instrumental activities of daily living such as preparing balanced meals and managing personal finances. The intent of the FAS is to assess change in an individual's functional activities, relative to previously attained abilities, that are caused by cognitive dysfunction. If the study partner indicates that the subject no longer performs a particular task, it is reasonable to probe further and ask if they think the subject could still do the task. This will help tease out the relevant cognitive impairment
  Scores range from 0-30 with lower scores indicate more favorable cognitive performance
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
units on a scale
  Week 52: number analyzed (Participants) | 43 | 36
  Week 52 | 0.68 (0.430) | 1.40 (0.469)
  Week 104: number analyzed (Participants) | 42 | 31
  Week 104 | 2.21 (0.690) | 2.44 (0.790)
  Week 156: number analyzed (Participants) | 38 | 29
  Week 156 | 3.03 (0.926) | 4.07 (1.061)
  Week 208: number analyzed (Participants) | 35 | 27
  Week 208 | 4.33 (1.208) | 5.55 (1.373)
  Week 260: number analyzed (Participants) | 12 | 7
  Week 260 | 5.82 (1.748) | 5.69 (2.073)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.507, t-test, 2 sided; Mean Difference (Final Values) = -1.22, 95% CI 2-sided [-4.86 to 2.42], Standard Error of Mean 1.828

10. Secondary Outcome: Solanezumab: Clinical Measures- Mini-Mental Status State Examination (MMSE)
Description: MMSE is a brief, quantitative measure of cognitive status in adults used to screen for cognitive impairment, to estimate the severity of cognitive impairment at a given point in time, to follow the course of cognitive changes in an individual over time, and to document an individual's response to treatment.
  Scores range from 0-30 and higher scores indicate more favorable cognitive function.
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
units on a scale
  Week 52: number analyzed (Participants) | 49 | 40
  Week 52 | -1.30 (0.354) | -0.83 (0.391)
  Week 104: number analyzed (Participants) | 47 | 36
  Week 104 | -2.59 (0.603) | -1.73 (0.677)
  Week 156: number analyzed (Participants) | 40 | 32
  Week 156 | -3.76 (0.858) | -3.23 (0.964)
  Week 208: number analyzed (Participants) | 36 | 30
  Week 208 | -5.31 (1.137) | -4.30 (1.275)
  Week 260: number analyzed (Participants) | 13 | 7
  Week 260 | -7.88 (1.799) | -5.94 (2.143)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.553, t-test, 2 sided; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-4.41 to 2.38], Standard Error of Mean 1.706

11. Secondary Outcome: Solanezumab: Cognitive Measures- International Shopping List Task 30-Minute Delayed Recall
Description: Classic list-learning test that measures verbal learning & memory.
  Scores range from 0-12 with higher scores indicating more favorable cognitive performance.
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
units on a scale
  Week 52: number analyzed (Participants) | 47 | 40
  Week 52 | -0.35 (0.248) | -0.17 (0.274)
  Week 104: number analyzed (Participants) | 47 | 35
  Week 104 | -0.98 (0.300) | -0.64 (0.343)
  Week 156: number analyzed (Participants) | 40 | 31
  Week 156 | -1.55 (0.294) | -0.42 (0.333)
  Week 208: number analyzed (Participants) | 35 | 28
  Week 208 | -1.92 (0.396) | -0.93 (0.447)
  Week 260: number analyzed (Participants) | 12 | 7
  Week 260 | -1.45 (0.548) | -1.86 (0.680)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.098, t-test, 2 sided; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-2.18 to 0.19], Standard Error of Mean 0.596

12. Secondary Outcome: Solanezumab: Cognitive Measures- Groton Maze Learning Test 30 Minute Delayed Recall
Description: The Groton Maze Learning Test 30 minute delayed recall measures episodic memory. The primary outcome is the number of errors made during recall of the previously memorized pathway from the Groton Maze Learning Test. The minimum score is 0 errors and the max is 999. Lower scores indicate better cognitive performance.
Time Frame: Baseline, Week 52, 104, 156, 208 and 260
Population: Number analyzed represents actual data collections at each collection time point. Data unavailable at any time point was not collected for various reasons i.e. participant attrition or common close design (participants did not reach that time point before trial end). Tasks are only included where assessed for subjects with a baseline Clinical Dementia Rating Global Score less than 1.
Measure: Least Squares Mean (Standard Error); unit: count of errors
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
count of errors
  Week 52: number analyzed (Participants) | 40 | 36
  Week 52 | 1.00 (0.975) | -0.13 (1.043)
  Week 104: number analyzed (Participants) | 37 | 31
  Week 104 | 1.16 (1.108) | 0.78 (1.207)
  Week 156: number analyzed (Participants) | 35 | 27
  Week 156 | 2.40 (1.055) | 0.96 (1.181)
  Week 208: number analyzed (Participants) | 32 | 24
  Week 208 | 4.33 (1.319) | 1.60 (1.470)
  Week 260: number analyzed (Participants) | 12 | 6
  Week 260 | 5.11 (2.894) | 6.99 (3.861)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.173, t-test, 2 sided; Mean Difference (Final Values) = 2.73, 95% CI 2-sided [-1.22 to 6.68], Standard Error of Mean 1.980

13. Secondary Outcome: Solanezumab: Cognitive Measures- Groton Maze Learning Test Delayed Reversed Recall
Description: The Groton Maze Learning Test measures executive function using a maze learning paradigm. A 10 x 10 grid of tiles is presented to the participant on the screen. A 28-step pathway is hidden among these tiles. A blue tile indicates the start and a tile with red circles indicates the finish. The participant must move one step at a time from the start toward the end by touching a tile next to their current location. If the correct move is made a green checkmark appears and if the move is incorrect a red cross is revealed. Once completed, they are returned to the start location to repeat the test and must try to remember the pathway they have just completed. "Delayed Reverse Recall" measures spatial working memory.
  The outcome is the number of errors made with the range of 0-999. Lower scores indicate better cognitive performance.
Time Frame: Baseline, Week 52, 104, 156, 208 and 260
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: number of errors
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
number of errors
  Week 52: number analyzed (Participants) | 40 | 36
  Week 52 | 7.08 (2.686) | -1.34 (2.858)
  Week 104: number analyzed (Participants) | 37 | 31
  Week 104 | 6.21 (2.715) | 3.28 (2.912)
  Week 156: number analyzed (Participants) | 35 | 28
  Week 156 | 6.45 (2.490) | 1.82 (2.711)
  Week 208: number analyzed (Participants) | 32 | 24
  Week 208 | 5.59 (2.658) | 5.29 (2.980)
  Week 260: number analyzed (Participants) | 12 | 6
  Week 260 | 14.25 (10.722) | 6.75 (15.509)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.940, t-test, 2 sided; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-8.10 to 8.71], Standard Error of Mean 3.998

14. Secondary Outcome: Solanezumab: Cognitive Measures- Trailmaking Test Part A
Description: Trail Making test taps attention, processing speed, and executive function. Part A consists of 25 circles numbered 1 through 25 distributed over a white sheet of standard document-sized paper. The subject is instructed to connect the circles with a drawn line as quickly as possible in ascending numerical order without lifting their pen.
  The subject's performance is judged in terms of the time, in seconds, required to complete each trail (Max time 150 seconds). Lower scores indicate more favorable cognitive function.
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
seconds
  Week 52: number analyzed (Participants) | 49 | 40
  Week 52 | 9.73 (2.895) | 5.14 (3.227)
  Week 104: number analyzed (Participants) | 45 | 33
  Week 104 | 15.03 (4.473) | 11.38 (5.039)
  Week 156: number analyzed (Participants) | 35 | 28
  Week 156 | 19.45 (5.832) | 15.21 (6.538)
  Week 208: number analyzed (Participants) | 33 | 25
  Week 208 | 35.69 (11.028) | 32.63 (12.430)
  Week 260: number analyzed (Participants) | 13 | 6
  Week 260 | 93.49 (27.664) | 89.02 (32.699)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.854, t-test, 2 sided; Mean Difference (Final Values) = 3.07, 95% CI 2-sided [-30.49 to 36.62], Standard Error of Mean 16.524

15. Secondary Outcome: Solanezumab: Cognitive Measures- Trailmaking Test Part B
Description: This test taps attention, processing speed, and executive function and depends on visuo-motor and perceptual-scanning skills and also requires considerable cognitive flexibility in shifting from number to letter sets under time pressure. Part B consists of 25 circles, but these circles contain either numbers (1 through 13) or letters (A through L). The subject must connect the circles while alternating between numbers and letters in an ascending order (e.g., A to 1; 1 to B; B to 2; 2 to C).
  The subject's performance is judged in terms of the time, in seconds, required to complete each Trail (Max of 300 seconds). Lower scores indicate more favorable cognitive function.
Time Frame: Baseline, Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: number of seconds
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
number of seconds
  Week 52: number analyzed (Participants) | 41 | 33
  Week 52 | -2.39 (6.582) | 8.00 (7.371)
  Week 104: number analyzed (Participants) | 36 | 27
  Week 104 | -0.20 (7.626) | 10.52 (8.710)
  Week 156: number analyzed (Participants) | 33 | 23
  Week 156 | 21.59 (11.619) | 21.35 (13.470)
  Week 208: number analyzed (Participants) | 29 | 23
  Week 208 | 21.42 (11.539) | 16.54 (13.211)
  Week 260: number analyzed (Participants) | 12 | 5
  Week 260 | 53.44 (25.139) | 37.62 (33.565)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.781, t-test, 2 sided; Mean Difference (Final Values) = 4.88, 95% CI 2-sided [-30.00 to 39.75], Standard Error of Mean 17.448

16. Secondary Outcome: Solanezumab: Cognitive Measures- WAIS-R Digit-Symbol Substitution Test
Description: This test engages multiple cognitive abilities, including attention, psychomotor speed, complex scanning, visual tracking, and immediate memory.
  Scores range from 0-93 with higher scores indicate more favorable cognitive function.
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
units on a scale
  Week 52: number analyzed (Participants) | 49 | 39
  Week 52 | 0.35 (1.149) | -1.02 (1.283)
  Week 104: number analyzed (Participants) | 41 | 32
  Week 104 | -0.97 (1.744) | 0.20 (1.965)
  Week 156: number analyzed (Participants) | 34 | 26
  Week 156 | -3.64 (2.232) | -1.72 (2.540)
  Week 208: number analyzed (Participants) | 33 | 26
  Week 208 | -7.83 (2.784) | -6.15 (3.170)
  Week 260: number analyzed (Participants) | 13 | 6
  Week 260 | -12.96 (4.057) | -9.60 (4.898)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.689, t-test, 2 sided; Mean Difference (Final Values) = -1.69, 95% CI 2-sided [-10.05 to 6.67], Standard Error of Mean 4.210

17. Secondary Outcome: Solanezumab: Cognitive Measures- WMS-R Digit Span Backward
Description: Widely used measure of working memory (or attention) in which the subject is read number sequences of increasing length and then asked to repeat each sequence backward. The primary measure of performance is the number of digit sequences correctly reversed.
  The unit of measure is number of digit sequences correctly recalled and ranges from 0-12. Higher scores indicate more favorable cognitive function.
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: number of correct sequences recalled
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
number of correct sequences recalled
  Week 52: number analyzed (Participants) | 49 | 40
  Week 52 | 0.06 (0.241) | -0.12 (0.267)
  Week 104: number analyzed (Participants) | 47 | 35
  Week 104 | -0.41 (0.272) | -0.16 (0.310)
  Week 156: number analyzed (Participants) | 40 | 32
  Week 156 | -1.14 (0.370) | -0.28 (0.415)
  Week 208: number analyzed (Participants) | 34 | 28
  Week 208 | -1.17 (0.460) | -0.68 (0.513)
  Week 260: number analyzed (Participants) | 12 | 6
  Week 260 | -1.17 (0.657) | -1.22 (0.832)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.474, t-test, 2 sided; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-1.86 to 0.87], Standard Error of Mean 0.689

18. Secondary Outcome: Solanezumab: Cognitive Measures- WMS-R Digit Span Forward
Description: This is a widely-used test of working memory in which the subject is read number sequences of increasing length and asked to repeat them. The total score is the number of sequences correctly repeated.
  The unit of measure is number of digit sequences correctly recalled and ranges from 0-12. Higher scores indicate more favorable cognitive function.
Time Frame: Baseline, Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: number of correct sequences recalled
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
number of correct sequences recalled
  Week 52: number analyzed (Participants) | 49 | 40
  Week 52 | -0.76 (0.220) | -0.38 (0.242)
  Week 104: number analyzed (Participants) | 47 | 35
  Week 104 | -1.03 (0.290) | -0.84 (0.329)
  Week 156: number analyzed (Participants) | 40 | 32
  Week 156 | -1.50 (0.346) | -1.23 (0.387)
  Week 208: number analyzed (Participants) | 35 | 28
  Week 208 | -1.96 (0.424) | -1.86 (0.475)
  Week 260: number analyzed (Participants) | 13 | 6
  Week 260 | -2.05 (0.722) | -1.06 (0.929)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.886, t-test, 2 sided; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-1.36 to 1.17], Standard Error of Mean 0.637

19. Secondary Outcome: Solanezumab: Cognitive Measures- Raven's Progressive Matrices (Set A)
Description: This is a measure of fluid intelligence. This test is used to get an estimate of the subjects IQ at baseline. Subjects are asked to complete a visual pattern by circling one of six response choices.
  Scores range from 0-12 with higher scores indicating more favorable cognitive performance.
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
units on a scale
  Week 52: number analyzed (Participants) | 49 | 39
  Week 52 | -0.47 (0.235) | -0.70 (0.261)
  Week 104: number analyzed (Participants) | 46 | 34
  Week 104 | -0.93 (0.310) | -0.63 (0.350)
  Week 156: number analyzed (Participants) | 38 | 31
  Week 156 | -1.38 (0.366) | -1.06 (0.408)
  Week 208: number analyzed (Participants) | 34 | 27
  Week 208 | -1.44 (0.372) | -1.53 (0.416)
  Week 260: number analyzed (Participants) | 13 | 6
  Week 260 | -3.11 (0.873) | -1.78 (1.124)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.873, t-test, 2 sided; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-1.03 to 1.20], Standard Error of Mean 0.556

20. Secondary Outcome: Solanezumab: Cognitive Measures- Category Fluency (Animals)
Description: Category Fluency is a widely used measure of semantic memory (verbal fluency, language). The subject is asked to name different exemplars of a given semantic category (animals), and the number of unique exemplars named is scored.
  Higher scores indicate more favorable cognitive function.
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
units on a scale
  Week 52: number analyzed (Participants) | 49 | 40
  Week 52 | -1.86 (0.642) | -2.19 (0.711)
  Week 104: number analyzed (Participants) | 47 | 35
  Week 104 | -1.64 (0.754) | -2.50 (0.860)
  Week 156: number analyzed (Participants) | 40 | 32
  Week 156 | -2.84 (0.869) | -2.46 (0.974)
  Week 208: number analyzed (Participants) | 35 | 28
  Week 208 | -4.69 (1.105) | -3.27 (1.239)
  Week 260: number analyzed (Participants) | 13 | 6
  Week 260 | -5.45 (1.761) | -6.50 (2.303)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.394, t-test, 2 sided; Mean Difference (Final Values) = -1.42, 95% CI 2-sided [-4.71 to 1.87], Standard Error of Mean 1.660

21. Secondary Outcome: Solanezumab: Cognitive Measures- Category Fluency (Vegetables)
Description: Category Fluency is a widely used measure of semantic memory (verbal fluency, language). The subject is asked to name different exemplars of a given semantic category (vegetables), and the number of unique exemplars named is scored.
  Higher scores indicate more favorable cognitive function.
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
units on a scale
  Week 52: number analyzed (Participants) | 49 | 40
  Week 52 | -0.83 (0.481) | -1.41 (0.533)
  Week 104: number analyzed (Participants) | 47 | 35
  Week 104 | -1.22 (0.539) | -1.74 (0.619)
  Week 156: number analyzed (Participants) | 40 | 32
  Week 156 | -1.29 (0.555) | -1.43 (0.623)
  Week 208: number analyzed (Participants) | 35 | 28
  Week 208 | -2.03 (0.707) | -1.72 (0.794)
  Week 260: number analyzed (Participants) | 13 | 6
  Week 260 | -3.36 (1.069) | -2.23 (1.386)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.776, t-test, 2 sided; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-2.41 to 1.81], Standard Error of Mean 1.063

22. Secondary Outcome: Solanezumab: Cognitive Measures- WMS-R Logical Memory Delayed Recall Test
Description: Measure of delayed recall (episodic memory) of a story read to the subject at the beginning of the testing session and subject is asked to relay the story 20 minutes later.
  Scores range from 0-25 with higher scores indicating more favorable cognitive performance.
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Pooled Placebo: Placebos enrolled under each arm but pooled for result reporting.
Arm/Group | Solanezumab | Pooled Placebo
Number analyzed (Participants) | 50 | 40
units on a scale
  Week 52: number analyzed (Participants) | 49 | 40
  Week 52 | 0.64 (0.397) | 1.33 (0.441)
  Week 104: number analyzed (Participants) | 47 | 34
  Week 104 | 1.25 (0.501) | 1.71 (0.576)
  Week 156: number analyzed (Participants) | 41 | 32
  Week 156 | 1.21 (0.549) | 2.37 (0.618)
  Week 208: number analyzed (Participants) | 35 | 28
  Week 208 | 0.84 (0.606) | 1.82 (0.678)
  Week 260: number analyzed (Participants) | 13 | 6
  Week 260 | 0.40 (1.029) | 2.68 (1.416)
Statistical Analysis 1: Comparison: Solanezumab vs Pooled Placebo; Test type: Other — Test of equality (any treatment difference); p = 0.283, t-test, 2 sided; Mean Difference (Final Values) = -0.98, 95% CI 2-sided [-2.78 to 0.82], Standard Error of Mean 0.909

23. Secondary Outcome: Solanezumab: Cognitive Measures- WMS-R Logical Memory Immediate Recall Test
Description: This test assesses the ability to recall a short story. The subject is read a short story and immediately after hearing the story, the subject is asked to retell the story from memory.
  Scores range from 0-25 with higher scores indicating more favorable cognitive performance.
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
units on a scale
  Week 52: number analyzed (Participants) | 49 | 40
  Week 52 | 0.40 (0.452) | -0.06 (0.501)
  Week 104: number analyzed (Participants) | 47 | 35
  Week 104 | 0.73 (0.510) | 0.75 (0.579)
  Week 156: number analyzed (Participants) | 41 | 32
  Week 156 | 0.13 (0.573) | 0.91 (0.646)
  Week 208: number analyzed (Participants) | 35 | 28
  Week 208 | 0.24 (0.631) | 0.69 (0.707)
  Week 260: number analyzed (Participants) | 13 | 6
  Week 260 | -0.56 (1.018) | 1.37 (1.420)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.634, t-test, 2 sided; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-2.33 to 1.42], Standard Error of Mean 0.947

24. Secondary Outcome: Solanezumab: Cognitive Measures- Composite Including: Alternative Multivariate Composite: (1) Digit Span Backwards; (2) Logical Memory (Immediate); (3) Trailmaking B; (4) Category Fluency (Animals)
Description: Multivariate Disease Progression Model adjusted for estimated years from symptom onset (EYO) and includes all time points up to treatment discontinuation. The treatment effect for Solanezumab is reported relative to the mutation positive placebo arm.
  This alternative multivariate endpoint includes four tests: Logical Memory Immediate Recall, Digit Span Backward Recall, Category Fluency (Animals), Trailmaking Test Part B. Measurements for each test will be normalized using the mean (SD) at DIAN-TU-001 baseline among mutation negative subjects before being analyzed. For the Trailmaking Test B, the scores will be multiplied by -1 as higher scores indicate worse performance; whereas for the other three, lower scores indicate worse performance. Therefore, on the standardized endpoints, lower scores indicate worse performance.
Time Frame: Baseline through Week 260
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Solanezumab vs. Mutation Positive Placebo Plus DIAN-OBS Control Group: Solanezumab: Intravenous infusion every 4 weeks at escalating doses; Matching Placebo
Arm/Group | Solanezumab vs. Mutation Positive Placebo Plus DIAN-OBS Control Group
Number analyzed (Participants) | 160
Ratio | 1.155 (0.074)
Statistical Analysis 1: Comparison: Solanezumab vs. Mutation Positive Placebo Plus DIAN-OBS Control Group; Test type: Superiority; A priori threshold for statistical significance; Ratio = 1.155, Standard Deviation 0.074

25. Secondary Outcome: Solanezumab: Imaging Measures- Brain Amyloid Load as Measured by [11C]PiB-PET Non-partial Volume Corrected
Description: PiB Standardized Uptake Value Ratio ([11C]PiB SUVR) is the most common quantitative method used to make regional comparisons within a subject as well as between subjects and computed as the degree of radiotracer uptake in a target region of interest (regions dervived via automated segmentation using FreeSurfer) with respect to a reference region. In amyloid and tau imaging, SUVR is typically generated using some portion or the entire cerebellum as a reference because cerebellum is not affected until late in the progression of AD.
Time Frame: Baseline and Weeks 52, 104 and 208
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
Ratio
  Week 52: number analyzed (Participants) | 46 | 37
  Week 52 | 0.030 (0.0147) | 0.025 (0.0164)
  Week 104: number analyzed (Participants) | 41 | 33
  Week 104 | 0.019 (0.0180) | 0.022 (0.0200)
  Week 208: number analyzed (Participants) | 27 | 25
  Week 208 | 0.113 (0.0387) | 0.093 (0.0408)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.726, t-test, 2 sided; Mean Difference (Final Values) = 0.020, 95% CI 2-sided [-0.093 to 0.132], Standard Error of Mean 0.0562

26. Secondary Outcome: Solanezumab: Imaging Measures- Brain Amyloid Load as Measured by Florbetapir PET
Description: Florbetapir Standardized Uptake Value Ratio ([18F]AV-45 SUVR) is the most common quantitative method used to make regional comparisons within a subject as well as between subjects and computed as the degree of radiotracer uptake in a target region of interest (regions derivved via automated segmentation using FreeSurfer) with respect to a reference region. In amyloid and tau imaging, SUVR is typically generated using some portion or the entire cerebellum as a reference because cerebellum is not affected until late in the progression of AD.
Time Frame: Weeks104 and 208
Population: Number analyzed represents actual data collections at each collection time point. Data unavailable at any time point was notcollected for various reasons i.e. participant attrition or common close design (participants did not reach that time point before trial end).
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
Ratio
  Week 104: number analyzed (Participants) | 36 | 29
  Week 104 | 0.066 (0.0458) | 0.105 (0.0511)
  Week 208: number analyzed (Participants) | 28 | 24
  Week 208 | 0.251 (0.0717) | 0.168 (0.0775)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.439, t-test, 2 sided; Mean Difference (Final Values) = 0.082, 95% CI 2-sided [-0.130 to 0.295], Standard Error of Mean 0.1056

27. Secondary Outcome: Solanezumab: Imaging Measures- Brain Glucose Metabolism as Measured by Fluorodeoxyglucose (FDG)-PET Non-partial Volume Corrected
Description: FDG Standardized Uptake Value Ratio ([18F]FDG SUVR) is the most common quantitative method used to make regional comparisons within a subject as well as between subjects and computed as the degree of radiotracer uptake in a target region of interest (regions derivved via automated segmentation using FreeSurfer) with respect to a reference region. In amyloid and tau imaging, SUVR is typically generated using some portion or the entire cerebellum as a reference because cerebellum is not affected until late in the progression of AD.
Time Frame: Baseline and Weeks 52, 104 and 208
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
Ratio
  Week 52: number analyzed (Participants) | 43 | 33
  Week 52 | -0.021 (0.0072) | -0.030 (0.0083)
  Week 104: number analyzed (Participants) | 42 | 31
  Week 104 | -0.047 (0.0063) | -0.043 (0.0074)
  Week 208: number analyzed (Participants) | 31 | 23
  Week 208 | -0.074 (0.0110) | -0.074 (0.0127)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.967, t-test, 2 sided; Mean Difference (Final Values) = 0.001, 95% CI 2-sided [-0.034 to 0.033], Standard Error of Mean 0.0168

28. Secondary Outcome: Solanezumab: Imaging Measures- Brain Atrophy as Measured by Cortical Thickness of Regions of Interest - Precuneus Region
Description: Brain atrophy was defined by structural magnetic resonance imaging (MRI) A Magnetization Prepared - RApid Gradient Echo) (MPRAGE) sequence was processed using the Freesurfer software suite. This package provides volumes and thickness values for cortical regions and volumes for subcortical regions. For the clinical trial we examined cortical thickness values in prespecified regions of interest known to show atrophy in autosomal dominant Alzheimer Disease. Higher measurements are more favorable.
Time Frame: Baseline and Weeks 52, 104, 156 and 208
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Millimeters
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
Millimeters
  Week 52: number analyzed (Participants) | 46 | 38
  Week 52 | -0.033 (0.0106) | -0.053 (0.0114)
  Week 104: number analyzed (Participants) | 43 | 35
  Week 104 | -0.067 (0.0142) | -0.090 (0.0156)
  Week 156: number analyzed (Participants) | 36 | 29
  Week 156 | -0.110 (0.0193) | -0.122 (0.0214)
  Week 208: number analyzed (Participants) | 32 | 28
  Week 208 | -0.138 (0.0254) | -0.154 (0.0279)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.669, t-test, 2 sided; Mean Difference (Final Values) = 0.016, 95% CI 2-sided [-0.059 to 0.092], Standard Error of Mean 0.0377

29. Secondary Outcome: Solanezumab: Imaging Measures- Volumetric MRI Combined Total Volume Corrected for Head Size - Hippocampus Volume
Description: Brain atrophy was defined by structural magnetic resonance imaging (MRI) A Magnetization Prepared - RApid Gradient Echo) (MPRAGE) sequence was processed using the Freesurfer software suite. This package provides volumes and thickness values for cortical regions and volumes for subcortical regions. For the clinical trial we examined volume values in prespecified regions of interest known to show atrophy in autosomal dominant Alzheimer Disease.
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Cubic Millimeters
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
Cubic Millimeters
  Week 52: number analyzed (Participants) | 46 | 38
  Week 52 | -106.74 (71.081) | -153.34 (78.529)
  Week 104: number analyzed (Participants) | 43 | 35
  Week 104 | -341.35 (72.549) | -302.58 (80.556)
  Week 156: number analyzed (Participants) | 36 | 29
  Week 156 | -524.14 (76.210) | -541.76 (84.861)
  Week 208: number analyzed (Participants) | 32 | 28
  Week 208 | -706.41 (78.746) | -671.95 (85.672)
  Week 260: number analyzed (Participants) | 10 | 7
  Week 260 | -977.91 (116.633) | -551.42 (137.366)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.768, t-test, 2 sided; Mean Difference (Final Values) = -34.46, 95% CI 2-sided [-264.14 to 195.22], Standard Error of Mean 116.419

30. Secondary Outcome: Solanezumab: Imaging Measures- Brain Tau Load as Measured by Flortaucipir PET Non-partial Volume Corrected
Description: This variable represents how much neurofibrillary tau pathology is present in brain as assessed using positron emission tomography (PET). Scans were conducted using [F18] Flortaucipir, a commonly used tracer in the field.
Time Frame: Baseline and Weeks 52, 104 and 208
Population: Number analyzed represents actual data collections at each collection time point. Data unavailable at any time point was not collected for various reasons i.e. participant attrition or common close design (participants did not reach that time point before trial end). In addition, the tau tracer was not introduced in the trial until after baseline for most participants.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
Ratio
  Baseline: number analyzed (Participants) | 7 | 6
  Baseline | 1.77391 (0.548324) | 1.52502 (0.582485)
  Week 52: number analyzed (Participants) | 21 | 19
  Week 52 | 1.46020 (0.503595) | 1.49041 (0.434475)
  Change in Baseline in Week 52: number analyzed (Participants) | 6 | 6
  Change in Baseline in Week 52 | 0.11302 (0.221413) | -0.03925 (0.192448)
  Week 104: number analyzed (Participants) | 28 | 21
  Week 104 | 1.49990 (0.506423) | 1.42231 (0.394000)
  Change from Baseline Week 104: number analyzed (Participants) | 6 | 4
  Change from Baseline Week 104 | 0.15450 (0.252682) | 0.01208 (0.263170)
  Week 208: number analyzed (Participants) | 19 | 12
  Week 208 | 1.43263 (0.402563) | 1.28081 (0.295191)
  Change from Baseline Week 208: number analyzed (Participants) | 2 | 2
  Change from Baseline Week 208 | 0.05275 (0.052679) | 0.05825 (0.023688)

31. Secondary Outcome: Solanezumab: Imaging Measures- Brain Atrophy as Measured by Whole Brain Volume Corrected for Head Size
Description: Brain atrophy was defined by structural magnetic resonance imaging (MRI) A Magnetization Prepared - RApid Gradient Echo) (MPRAGE) sequence was processed using the Freesurfer software suite. This package provides volumes and thickness values for cortical regions and volumes for subcortical regions. A whole brain volume measure was generated to represent global atrophy across the cortical and subcortical regions.
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Cubic Millimeters
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
Cubic Millimeters
  Week 52: number analyzed (Participants) | 46 | 38
  Week 52 | -11990.31 (4027.589) | -10578.56 (4409.442)
  Week 104: number analyzed (Participants) | 43 | 35
  Week 104 | -19808.05 (4106.838) | -22147.27 (4524.072)
  Week 156: number analyzed (Participants) | 36 | 29
  Week 156 | -32713.22 (4304.849) | -30590.95 (4770.402)
  Week 208: number analyzed (Participants) | 32 | 28
  Week 208 | -39306.90 (4446.803) | -36569.28 (4816.319)
  Week 260: number analyzed (Participants) | 10 | 7
  Week 260 | -54558.23 (6562.583) | -50077.53 (7713.907)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.677, t-test, 2 sided; Mean Difference (Final Values) = -2737.62, 95% CI 2-sided [-15678.06 to 10202.81], Standard Error of Mean 6558.467

32. Secondary Outcome: Solanezumab: Imaging Measures- Brain Atrophy as Measured by Ventricular Volume (Volumetric MRI) Corrected for Head Size
Description: Rather than looking at how tissue in the brain changes, it is also possible to quantify how the ventricles, fluid filled spaces in the brain, change. Increasing ventricular volume represents greater amounts of cerebral spinal fluid which suggests atrophy of the brain. Magnetization Prepared - RApid Gradient Echo) (MPRAGE) sequences were processed using the Freesurfer software suite. Total ventricular volume was calculated from the ventricular volumes generated by this program.
Time Frame: Baseline and Weeks 52, 104, 156, 208 and 260
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Cubic Millimeters
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
Cubic Millimeters
  Week 52: number analyzed (Participants) | 46 | 38
  Week 52 | 1815.99 (1067.526) | 1796.78 (1182.631)
  Week 104: number analyzed (Participants) | 43 | 35
  Week 104 | 2972.85 (1094.409) | 4452.69 (1218.440)
  Week 156: number analyzed (Participants) | 36 | 29
  Week 156 | 5705.59 (1163.978) | 6729.64 (1297.406)
  Week 208: number analyzed (Participants) | 32 | 28
  Week 208 | 8755.04 (1212.184) | 9833.37 (1312.937)
  Week 260: number analyzed (Participants) | 10 | 7
  Week 260 | 12332.3 (1907.752) | 11456.61 (2258.240)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.547, t-test, 2 sided; Mean Difference (Final Values) = -1078.32, 95% CI 2-sided [-4603.28 to 2446.64], Standard Error of Mean 1788.474

33. Secondary Outcome: Solanezumab: Fluid Biomarker Measures- CSF Aβ 40 Free Change From Baseline
Description: Measured concentration of the drug bound and free soluble Aβ1-40 peptide in cerebrospinal fluid using enzyme-linked immunosorbent assay (ELISA)
Time Frame: Baseline and Weeks 52, 104 and 208
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Groups:
- Solanezumab Direct Placebo: Subjects enrolled under solanezumab placebo arm
Arm/Group | Solanezumab | Solanezumab Direct Placebo
Number analyzed (Participants) | 50 | 19
pg/mL
  Week 52: number analyzed (Participants) | 41 | 18
  Week 52 | -1613.48 (185.134) | -856.65 (284.584)
  Week 104: number analyzed (Participants) | 42 | 15
  Week 104 | -2237.73 (177.616) | -1398.13 (290.994)
  Week 208: number analyzed (Participants) | 24 | 13
  Week 208 | -2567.13 (229.807) | -631.22 (307.331)
Statistical Analysis 1: Comparison: Solanezumab vs Solanezumab Direct Placebo; Test type: Other — Test of equality (any treatment difference); p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -1935.91, 95% CI 2-sided [-2717.64 to -1154.18], Standard Error of Mean 385.538

34. Secondary Outcome: Solanezumab: Fluid Biomarker Measures- CSF Aβ 42 Free
Description: Measured concentration of the total soluble Aβ 1-42 peptide in cerebrospinal fluid using ELISA
Time Frame: Baseline and Weeks 52, 104 and 208
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Solanezumab | Solanezumab Direct Placebo
Number analyzed (Participants) | 50 | 19
pg/mL
  Week 52: number analyzed (Participants) | 40 | 17
  Week 52 | -109.33 (24.235) | -79.35 (37.602)
  Week 104: number analyzed (Participants) | 40 | 14
  Week 104 | -172.55 (14.535) | -125.64 (24.402)
  Week 208: number analyzed (Participants) | 19 | 11
  Week 208 | -250.78 (13.935) | -173.66 (18.204)
Statistical Analysis 1: Comparison: Solanezumab vs Solanezumab Direct Placebo; Test type: Other — Test of equality (any treatment difference); p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = -77.12, 95% CI 2-sided [-124.56 to -29.68], Standard Error of Mean 23.014

35. Secondary Outcome: Solanezumab: Fluid Biomarker Measures- CSF Tau
Description: Measured concentration of the soluble Tau peptide in cerebrospinal fluid
Time Frame: Baseline and Weeks 52, 104 and 208
Population: Number analyzed represents actual data collections at each collection time point. Data was not collected for all participants at each time point for various reasons
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
pg/mL
  Week 52: number analyzed (Participants) | 38 | 35
  Week 52 | 4.73 (14.884) | -6.60 (15.553)
  Week 104: number analyzed (Participants) | 38 | 32
  Week 104 | 31.74 (15.649) | 23.24 (16.783)
  Week 208: number analyzed (Participants) | 29 | 28
  Week 208 | 59.08 (24.691) | 28.19 (25.579)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.388, t-test, 2 sided; Mean Difference (Final Values) = 30.89, 95% CI 2-sided [-40.04 to 101.83], Standard Error of Mean 35.540

36. Secondary Outcome: Solanezumab: Fluid Biomarker Measures- CSF pTau 181
Description: Measured concentration of phosphorylated tau at threonine-181 in cerebrospinal fluid
Time Frame: Baseline and Weeks 52, 104 and 208
Population: as for outcome 35
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
pg/mL
  Week 52: number analyzed (Participants) | 45 | 37
  Week 52 | 0.26 (2.951) | -0.18 (3.254)
  Week 104: number analyzed (Participants) | 43 | 34
  Week 104 | 4.91 (2.903) | 4.25 (3.290)
  Week 208: number analyzed (Participants) | 32 | 29
  Week 208 | 6.90 (4.447) | 7.65 (4.907)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.909, t-test, 2 sided; Mean Difference (Final Values) = -0.76, 95% CI 2-sided [-13.97 to 12.45], Standard Error of Mean 6.624

37. Secondary Outcome: Solanezumab: Change From Baseline Fluid Biomarker Measures- CSF Neurofilament Light Chain (NfL)
Description: Measured concentration of neurofilament light chain in cerebrospinal fluid using SIMO
Time Frame: Baseline and Weeks 52, 104 and 208
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
pg/mL
  Week 52: number analyzed (Participants) | 44 | 35
  Week 52 | 0.102 (0.0414) | 0.144 (0.0463)
  Week 104: number analyzed (Participants) | 42 | 33
  Week 104 | 0.191 (0.0314) | 0.159 (0.0354)
  Week 208: number analyzed (Participants) | 31 | 28
  Week 208 | 0.426 (0.0402) | 0.248 (0.0435)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.004, t-test, 2 sided; Mean Difference (Final Values) = 0.178, 95% CI 2-sided [0.059 to 0.296], Standard Error of Mean 0.0593

38. Secondary Outcome: Solanezumab: Fluid Biomarker Measures- Plasma Neurofilament Light Chain (NfL)
Description: Measured concentration of neurofilamnet light chain in plasma using Single Molecule Array (SIMOA)
Time Frame: Baseline and Weeks 52, 104 and 208
Population: as for outcome 35
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 50 | 40
pg/mL
  Week 52: number analyzed (Participants) | 37 | 36
  Week 52 | 0.47 (1.864) | 4.03 (1.893)
  Week 104: number analyzed (Participants) | 32 | 33
  Week 104 | 1.22 (0.799) | 3.15 (0.780)
  Week 208: number analyzed (Participants) | 26 | 26
  Week 208 | 3.29 (0.959) | 3.72 (0.960)
Statistical Analysis 1: Comparison: Solanezumab vs Mutation Positive Placebos; Test type: Other — Test of equality (any treatment difference); p = 0.754, t-test, 2 sided; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-3.21 to 2.35], Standard Error of Mean 1.355

39. Secondary Outcome: Solanezumab: Fluid Biomarker Measures- Plasma Anti-drug Antibodies (ADA)
Description: Measurement of the presence or absence of anti-drug antibodies in serum
  Note: Mutation Negative Placebo subjects are not displayed as anti-drug antibody testing was not to be evaluated for these subjects.
  Note: Treatment Emergent Anti-Drug Antibody Positive subjects are defined as those with either (a) a baseline status of ADA Not Present and at least one post-baseline ADA present with a titer >= 1:20 or (b) both a baseline and post-baseline status of ADA Present with the post-baseline titer being 2 dilutions (4-fold) greater than the baseline titer.
  Note: Treatment Emergent Anti-Drug Antibody Inconclusive subjects are defined as those for whom >=20% of the subject's post-baseline ADA results are ADA Inconclusive and all remaining post-baseline samples are ADA Not Present.
  Note: Treatment Emergent Anti-Drug Antibody Negative subjects are defined as those who are evaluable for TE ADA but are neither TE ADA Positive nor TE ADA Inconclusive.
Time Frame: Baseline and Weeks 52, 104 and 208
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Solanezumab | Mutation Positive Placebos
Number analyzed (Participants) | 52 | 40
Participants
  Baseline : Not Detected: number analyzed (Participants) | 46 | 25
  Baseline : Not Detected | 43 | 22
  Baseline : Detected: number analyzed (Participants) | 46 | 25
  Baseline : Detected | 3 | 3
  Baseline: Detected Titer 1:10: number analyzed (Participants) | 46 | 25
  Baseline: Detected Titer 1:10 | 2 | 3
  Baseline: Detected Titer 1:20: number analyzed (Participants) | 46 | 25
  Baseline: Detected Titer 1:20 | 1 | 0
  Week 52 : Not Detected: number analyzed (Participants) | 48 | 35
  Week 52 : Not Detected | 44 | 32
  Week 52 : Detected: number analyzed (Participants) | 48 | 35
  Week 52 : Detected | 4 | 3
  Week 52 : Detected Titer 1:10: number analyzed (Participants) | 48 | 35
  Week 52 : Detected Titer 1:10 | 3 | 2
  Week 52 : Detected Titer 1:20: number analyzed (Participants) | 48 | 35
  Week 52 : Detected Titer 1:20 | 0 | 1
  Week 52 : Detected Titer 1:80: number analyzed (Participants) | 48 | 35
  Week 52 : Detected Titer 1:80 | 1 | 0
  Week 104 : Not Detected: number analyzed (Participants) | 43 | 32
  Week 104 : Not Detected | 40 | 29
  Week 104 : Detected: number analyzed (Participants) | 43 | 32
  Week 104 : Detected | 3 | 3
  Week 104 : Detected Titer 1:10: number analyzed (Participants) | 43 | 32
  Week 104 : Detected Titer 1:10 | 0 | 2
  Week 104 : Detected Titer 1:20: number analyzed (Participants) | 43 | 32
  Week 104 : Detected Titer 1:20 | 1 | 1
  Week 104 : Detected Titer 1:80: number analyzed (Participants) | 43 | 32
  Week 104 : Detected Titer 1:80 | 1 | 0
  Week 104 : Detected Titer 1:320: number analyzed (Participants) | 43 | 32
  Week 104 : Detected Titer 1:320 | 1 | 0
  Week 208 : Not Detected: number analyzed (Participants) | 35 | 26
  Week 208 : Not Detected | 33 | 24
  Week 208 : Detected: number analyzed (Participants) | 35 | 26
  Week 208 : Detected | 2 | 2
  Week 208 : Detected Titer 1:10: number analyzed (Participants) | 35 | 26
  Week 208 : Detected Titer 1:10 | 1 | 1
  Week 208 : Detected Titer 1:20: number analyzed (Participants) | 35 | 26
  Week 208 : Detected Titer 1:20 | 1 | 1
  Treatment Emergent ADA Positive: number analyzed (Participants) | 46 | 25
  Treatment Emergent ADA Positive | 2 | 0
  >=1 Positive Neutralizing Antibody Result: number analyzed (Participants) | 46 | 25
  >=1 Positive Neutralizing Antibody Result | 0 | 0
  Treatment Emergent ADA Inconclusive: number analyzed (Participants) | 46 | 25
  Treatment Emergent ADA Inconclusive | 0 | 0
  Treatment Emergent ADA Negative: number analyzed (Participants) | 46 | 25
  Treatment Emergent ADA Negative | 44 | 25

40. Secondary Outcome: Solanezumab: Fluid Biomarker Measures- Total Plasma Aβ 1-40
Description: Measured concentration of the total soluble Aβ 1-40 peptide in cerebrospinal fluid using ELISA
Time Frame: Baseline and Weeks 52, 104 and 208
Population: as for outcome 35
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Solanezumab | Solanezumab Direct Placebo
Number analyzed (Participants) | 50 | 19
pg/mL
  Week 52: number analyzed (Participants) | 45 | 19
  Week 52 | 168588.48 (5889.151) | -9257.53 (9091.376)
  Week 104: number analyzed (Participants) | 40 | 14
  Week 104 | 165220.34 (5425.379) | -9263.35 (9010.529)
  Week 208: number analyzed (Participants) | 31 | 14
  Week 208 | 220136.05 (8168.936) | -9226.25 (12358.817)
Statistical Analysis 1: Comparison: Solanezumab vs Solanezumab Direct Placebo; Test type: Other — Test of equality (any treatment difference); p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 229362.30, 95% CI 2-sided [199264.32 to 259460.27], Standard Error of Mean 14863.080

41. Secondary Outcome: Solanezumab: Fluid Biomarker Measures- Total Plasma Aβ 42
Description: Measured concentration of the total soluble Aβ 1-42 peptide in cerebrospinal fluid using ELISA
Time Frame: Baseline and Weeks 52, 104 and 208
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Solanezumab | Solanezumab Direct Placebo
Number analyzed (Participants) | 50 | 19
pg/mL
  Week 52: number analyzed (Participants) | 34 | 15
  Week 52 | 30609.39 (1555.170) | 526.91 (2334.054)
  Week 104: number analyzed (Participants) | 31 | 11
  Week 104 | 29265.35 (1459.112) | 746.90 (2424.659)
  Week 208: number analyzed (Participants) | 24 | 11
  Week 208 | 33744.89 (922.711) | 838.29 (1415.925)
Statistical Analysis 1: Comparison: Solanezumab vs Solanezumab Direct Placebo; Test type: Other — Test of equality (any treatment difference); p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 32906.60, 95% CI 2-sided [29406.49 to 36406.72], Standard Error of Mean 1697.541

42. Secondary Outcome: Solanezumab: Fluid Biomarker Measures- CSF Aβ 42 Total
Description: Measured concentration of the total soluble Aβ1-42 peptide in cerebrospinal fluid using enzyme-linked immunosorbent assay (ELISA)
Time Frame: Baseline and Weeks 52, 104 and 208
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Solanezumab | Solanezumab Direct Placebo
Number analyzed (Participants) | 50 | 19
pg/mL
  Week 52: number analyzed (Participants) | 39 | 17
  Week 52 | 558.91 (44.533) | 44.81 (69.142)
  Week 104: number analyzed (Participants) | 40 | 14
  Week 104 | 623.16 (41.301) | 89.32 (68.119)
  Week 208: number analyzed (Participants) | 27 | 12
  Week 208 | 1352.83 (75.447) | 66.48 (118.662)
Statistical Analysis 1: Comparison: Solanezumab vs Solanezumab Direct Placebo; Test type: Other — Test of equality (any treatment difference); p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 1286.35, 95% CI 2-sided [1002.79 to 1569.90], Standard Error of Mean 140.692

43. Secondary Outcome: Solanezumab: Fluid Biomarker Measures- CSF Aβ 40 Total
Description: Measured concentration of the total soluble Aβ1-40 peptide in cerebrospinal fluid using enzyme-linked immunosorbent assay (ELISA)
Time Frame: Baseline and Weeks 52, 104 and 208
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Solanezumab | Solanezumab Direct Placebo
Number analyzed (Participants) | 50 | 19
pg/mL
  Week 52: number analyzed (Participants) | 42 | 18
  Week 52 | 3676.97 (403.908) | -414.57 (625.000)
  Week 104: number analyzed (Participants) | 42 | 15
  Week 104 | 4017.93 (331.917) | -594.08 (549.240)
  Week 208: number analyzed (Participants) | 29 | 13
  Week 208 | 9723.95 (669.037) | -143.31 (1011.672)
Statistical Analysis 1: Comparison: Solanezumab vs Solanezumab Direct Placebo; Test type: Other — Test of equality (any treatment difference); p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 9867.26, 95% CI 2-sided [7419.38 to 12315.15], Standard Error of Mean 1212.232

ADVERSE EVENTS:
Time Frame: AE data was collected from consenting up to post study follow-up 8-12 weeks after last dose, approximately 6 years overall.
Description: In order to protect the genetic blinding requested by participants, as well as treatment assignment in the double-blind period to protect integrity of the ongoing open-label extension, the following precautions have been taken: 1) All Other (Not Including Serious) AEs have been reported by the higher level SOC; 2) SAEs have been summarized per arm at the general organ system level, and additionally at the subject level using a combined Arm/Group necessary to preserve participant confidentiality
Groups:
- Gantenerumab: Gantenerumab Active Treatment: Dosing subcutaneously every 4 weeks at escalating doses
- Solanezumab: Solanezumab Active Treatment: Dosing by intravenous infusion every 4 weeks at escalating doses
- Placebo: All placebos including mutation negative and positive
- DIAN OBS Control Group: Participants in the DIAN-OBS study who met DIAN-TU inclusion criteria were used as natural history controls for improved estimates of the placebo group.
  DIAN-OBS participants were included based on specific criteria as outlined in the SAP; included at the first visit where eligibility was met which means their period of eligibility would not match the full period of time as the DIAN-TU-001 placebo participants.
- Combined Blinded: All arms/groups combined for the purpose of maintaining blinding for participant mutation status and treatment group.
Arm/Group | Gantenerumab | Solanezumab | Placebo | DIAN OBS Control Group | Combined Blinded
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52 | 0/89 | 1/69 | 0/0
Serious Adverse Events (participants affected / at risk) | 12/52 | 13/52 | 12/89 | 10/69 | 47/262
Other Adverse Events (participants affected / at risk) | 52/52 | 52/52 | 89/89 | 57/69 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Gantenerumab (N=52) | Solanezumab (N=52) | Placebo (N=89) | DIAN OBS Control Group (N=69) | Combined Blinded (N=262)
General disorders (General disorders) | 12 (19) | 13 (17) | 12 (23) | 10 (11) | 0/0 (0) — To maintain blinding to participants' genetic status and assigned treatment, SAEs reported at the arm/group level are included under the General disorders SOC; all other SOCs are reported in the Combined Blinded Group.
Gastrointestinal disorders (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 7 (8) — To maintain blinding to participants' genetic status and assigned treatment, SAEs reported at the arm/group level are included under the General disorders SOC; all other SOCs are reported in the Combined Blinded Group.
General disorders (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 3 (3) — To maintain blinding to participants' genetic status and assigned treatment, SAEs reported at the arm/group level are included under the General disorders SOC; all other SOCs are reported in the Combined Blinded Group.
Infections and infestations (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 9 (9) — To maintain blinding to participants' genetic status and assigned treatment, SAEs reported at the arm/group level are included under the General disorders SOC; all other SOCs are reported in the Combined Blinded Group.
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 14 (16) — To maintain blinding to participants' genetic status and assigned treatment, SAEs reported at the arm/group level are included under the General disorders SOC; all other SOCs are reported in the Combined Blinded Group.
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 6 (6) — To maintain blinding to participants' genetic status and assigned treatment, SAEs reported at the arm/group level are included under the General disorders SOC; all other SOCs are reported in the Combined Blinded Group.
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 3 (3) — To maintain blinding to participants' genetic status and assigned treatment, SAEs reported at the arm/group level are included under the General disorders SOC; all other SOCs are reported in the Combined Blinded Group.
Nervous system disorders (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 11 (12) — To maintain blinding to participants' genetic status and assigned treatment, SAEs reported at the arm/group level are included under the General disorders SOC; all other SOCs are reported in the Combined Blinded Group.
Psychiatric disorders (Psychiatric disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 4 (4) — To maintain blinding to participants' genetic status and assigned treatment, SAEs reported at the arm/group level are included under the General disorders SOC; all other SOCs are reported in the Combined Blinded Group.
Renal and urinary disorders (Renal and urinary disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 3 (3) — To maintain blinding to participants' genetic status and assigned treatment, SAEs reported at the arm/group level are included under the General disorders SOC; all other SOCs are reported in the Combined Blinded Group.
Reproductive system and breast disorders (Reproductive system and breast disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 2 (2) — To maintain blinding to participants' genetic status and assigned treatment, SAEs reported at the arm/group level are included under the General disorders SOC; all other SOCs are reported in the Combined Blinded Group.
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 2 (2) — To maintain blinding to participants' genetic status and assigned treatment, SAEs reported at the arm/group level are included under the General disorders SOC; all other SOCs are reported in the Combined Blinded Group.
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 2 (2) — To maintain blinding to participants' genetic status and assigned treatment, SAEs reported at the arm/group level are included under the General disorders SOC; all other SOCs are reported in the Combined Blinded Group.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gantenerumab (N=52) | Solanezumab (N=52) | Placebo (N=89) | DIAN OBS Control Group (N=69) | Combined Blinded (N=0)
Cardiac Disorders (Cardiac disorders) | 4 (5) | 1 (2) | 9 (13) | 0 | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Ear and labyrinth disorders (Ear and labyrinth disorders) | 8 (8) | 6 (8) | 11 (17) | 0 | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Eye Disorders (Eye disorders) | 12 (18) | 2 (3) | 9 (11) | 0 | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Gastrointestinal disorders (Gastrointestinal disorders) | 33 (115) | 35 (88) | 48 (133) | 0 | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
General disorders and administration site conditions (General disorders) | 50 (1066) | 31 (70) | 54 (262) | 0 | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Immune system disorders (Immune system disorders) | 5 (6) | 8 (10) | 8 (9) | 0 | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 36 (92) | 35 (85) | 52 (146) | 27 (35) | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Investigations (Investigations) | 16 (31) | 12 (19) | 30 (55) | 0 | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 7 (11) | 6 (7) | 14 (17) | 0 | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 30 (95) | 28 (89) | 52 (140) | 25 (38) | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 5 (7) | 4 (5) | 0 | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Nervous system disorders (Nervous system disorders) | 41 (192) | 38 (175) | 58 (276) | 30 (48) | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Psychiatric disorders (Psychiatric disorders) | 22 (55) | 29 (51) | 29 (50) | 0 | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Renal and urinary disorders (Renal and urinary disorders) | 5 (6) | 4 (5) | 6 (7) | 0 | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Reproductive system and breast disorders (Reproductive system and breast disorders) | 7 (7) | 6 (7) | 8 (10) | 0 | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 24 (54) | 22 (64) | 33 (91) | 0 | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 23 (52) | 18 (36) | 29 (49) | 0 | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Vascular disorders (Vascular disorders) | 8 (10) | 5 (7) | 13 (18) | 0 | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Infections and infestations (Infections and infestations) | 39 (180) | 41 (170) | 62 (223) | 0 | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.
Social Circumstances (Social circumstances) | 3 (4) | 3 (3) | 5 (7) | 0 | NA — In order to maintain blinding to participants' genetic status and assigned treatment, this AE is reported by system organ class.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's may publish data and study results individually after the earlier of: 1) multi-center Publication is published; 2) no multi-center publication is submitted within 18 months after conclusion, abandonment, or termination of the Protocol at all sites; or 3) sponsor confirms in writing there will be no multi-center Publication. PI must submit results communications to the sponsor at least 75 days prior to submission or presentation. Sponsor can require changes to the communication.

DOCUMENTS (2):
  • Study Protocol (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT04623242/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT04623242/SAP_001.pdf